CLINICAL TRIAL: NCT03927703
Title: A Phase 3 Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study Comparing the Efficacy and Safety of SB206 and Vehicle Gel Once Daily in the Treatment of Molluscum Contagiosum
Brief Title: A Phase 3 Efficacy & Safety of SB206 & Vehicle Gel for the Treatment of MC
Acronym: B-SIMPLE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-MC302
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SB206 12% (Experimental): SB206 12% topically once daily
  Interventions: Drug: SB206 12%
- Placebo Comparator (Placebo Comparator): Placebo topically once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB206 12% — Topically once daily
  Other Names: berdazimer sodium
  Arms: SB206 12%
Drug: Placebo — Topically once daily
  Other Names: Vehicle Gel
  Arms: Placebo Comparator

SUMMARY:
This is a Phase 3 multi-center, randomized, double-blind, vehicle-controlled, parallel group study to be conducted in up to approximately 340 subjects ≥6 months of age with MC. Subjects or their caregivers will apply SB206 12% or Vehicle Gel once daily for a minimum of 4 weeks and up to 12 weeks to all lesions identified at Baseline and new treatable lesions that arise during the course of the study.

DETAILED DESCRIPTION:
This is a Phase 3 multi-center, randomized, double-blind, vehicle-controlled, parallel group study to be conducted in approximately 340 subjects with MC. After obtaining informed consent/assent, subjects who satisfy entry criteria will be randomized 2:1 (active:vehicle). Subjects receiving current treatment for MC at the time of the Screening Visit will enter a wash out period of up to 14 days prior to randomization.

Subjects or their caregivers will apply SB206 12% or Vehicle Gel once daily for a minimum of 4 weeks and up to 12 weeks to all lesions identified at Baseline and new treatable lesions that arise during the course of the study. Subjects or their caregivers will continue to treat the area until the next scheduled visit even if the lesion(s) clear. If the investigator determines all lesions are cleared at a clinic visit, the treatment may stop. Subjects will visit the clinic at Screening/Baseline, Week 2, Week 4, Week 8, Week 12. In addition, subjects will be seen in the clinic for a safety follow-up at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Be 6 months of age or older, and in good general health;
* Have a written informed consent form signed by subject or a parent or legal guardian and an assent form as required;
* Have between 3 and 70 treatable MC at Baseline;
* Female subjects age 9 and above must have a negative UPT at Baseline;
* Female subjects age 9 and above must agree to practice a medically acceptable form of birth control during the study and for 30 days after Week 12/ET1;
* Be willing and able to follow study instructions and likely to complete all study requirements.

Exclusion Criteria:

* Have strongly suggested sexually transmitted MC and do not agree to refrain from sexual activities throughout the study period.
* Are immunosuppressed, have immunodeficiency disorder, or are on immunosuppressive treatment;
* Have significant injury on and/or surrounding MC that may impact ability to treat and count lesions;
* Have received treatment with topical calcineurin inhibitors or steroids on MC or within 2 cm of MC lesions within 14 days prior to Baseline;
* Have received treatment for MC during the 14 days prior to Baseline with podophyllotoxin, imiquimod, cantharidin, sinecatechins, topical retinoids, oral or topical zinc, or other homeopathic or over the counter (OTC) products including, but not limited to, ZymaDerm and tea tree oil, cimetidine and other histamine H2 receptor antagonists (including Zantac);
* Have received surgical procedures related to MC (cryotherapy, curettage, other) within 14 days prior to Baseline;
* Have MC only in periocular area;
* Female subjects who are pregnant, planning a pregnancy or breastfeeding;
* Have known hypersensitivity to any ingredients of SB206 or Vehicle Gel including excipients;
* Have participated in a previous study with a berdazimer sodium product (SB204, SB206, SB208, SB414);
* Have more than 1 family member currently participating in a study with a berdazimer sodium product (SB204, SB206, SB208, SB414).
* Have participated in any other trial of an interventional investigational drug or device within 14 days or concurrent participation in another interventional research study.
* History or presence of clinically significant medical, psychiatric, or emotional condition that, in opinion of the investigator, would compromise the safety of the subject or the quality of the data.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adelaide Hebert, MD, Principal Investigator — UTHealth McGovern Medical School, Houston
Locations (27):
- United States (27):
  - Site #266, Scottsdale, Arizona
  - Site #101, Hot Springs, Arkansas
  - Site #282, Beverly Hills, California
  - Site #113, San Diego, California
  - Site #257, Thornton, Colorado
  - Site #268, Boynton Beach, Florida
  - Site #292, DeLand, Florida
  - Site #278, Miami, Florida
  - Site #305, Tampa, Florida
  - Site #175, New Albany, Indiana
  - Site #294, Owensboro, Kentucky
  - Site #289, Metairie, Louisiana
  - Site #297, New Orleans, Louisiana
  - Site #275, Largo, Maryland
  - Site #274, Clarkston, Michigan
  - Site #121, Fridley, Minnesota
  - Site #206, Omaha, Nebraska
  - Site #304, Portsmouth, New Hampshire
  - Site #201, Berlin, New Jersey
  - Site #108, Rochester, New York
  - Site #309, Portland, Oregon
  - Site #255, Mt. Pleasant, South Carolina
  - Site #271, Knoxville, Tennessee
  - Site #167, Houston, Texas
  - Site #293, Plano, Texas
  - Site #281, Syracuse, Utah
  - Site #267, Richmond, Virginia

REFERENCES:
- [Derived] Maeda-Chubachi T, Hebert D, Messersmith E, Siegfried EC. SB206, a Nitric Oxide-Releasing Topical Medication, Induces the Beginning of the End Sign and Molluscum Clearance. JID Innov. 2021 May 5;1(3):100019. doi: 10.1016/j.xjidi.2021.100019. eCollection 2021 Sep. PMID 34909721

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began June 13, 2019 and ended on August 12, 2019
Pre-assignment Details: Subjects receiving current treatment for MC at the time of the Screening Visit will enter a wash out period of up to 14 days prior to randomization.
Period: Overall Study
Arm/Group | SB206 12% | Placebo Comparator
Started | 237 | 118
Completed | 192 | 102
Not Completed | 45 | 16

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population--consisted of all subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | SB206 12% | Placebo Comparator | Total
Number analyzed (Participants) | 237 | 118 | 355
Age, Customized [Number; unit: participants]
  <1 year old | 0 | 0 | 355
  1 to 2 years old | 5 | 3 | 8
  2 years old to 6 years old | 116 | 60 | 176
  6 years old to 12 years old | 108 | 46 | 154
  12 years old to 18 years old | 8 | 7 | 15
  18 years old | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 62 | 172
  Male | 127 | 56 | 183
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 21 | 53
  Not Hispanic or Latino | 202 | 96 | 298
  Ethnicity Not Reported | 3 | 0 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Black or African American | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 221 | 104 | 325
  More than One Race | 3 | 6 | 9
  Race Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 237 | 117 | 354
Baseline number of Molluscum lesions [Mean (Standard Deviation); unit: Molluscum lesions] | 18.9 (14.46) | 17.1 (12.82) | 18.3 (13.95)

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance of All Treatable MC at Week 12
Description: Percent (proportion) of subjects with complete clearance of all treatable MC at Week 12. This was measured by dividing the number of subjects who showed complete clearance by the number in that treatment group (this represents our primary outcome variable).
Time Frame: 12 Weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- SB206: SB206 applied every day for 12 weeks.
- Placebo: Placebo gel applied every day for 12 weeks.
Arm/Group | SB206 | Placebo
Number analyzed (Participants) | 237 | 118
Participants | 71 | 24

2. Secondary Outcome: Complete Clearance of All Treatable MC at Week 8
Description: Percent (proportion) of subjects with complete clearance of all treatable MC at Week 8. This was measured by dividing the number of subjects who showed complete clearance at week 8 by the number in that treatment group (this represents our secondary outcome variable).
Time Frame: 8 Weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- SB206: SB206 gel applied once daily for 12 weeks.
- Placebo: Placebo gel applied once daily for 12 weeks.
Arm/Group | SB206 | Placebo
Number analyzed (Participants) | 237 | 118
Participants | 33 | 7

ADVERSE EVENTS:
Time Frame: Baseline visit to end of study visit, 84 days.
Description: Only TEAEs were to be considered. Adverse Events were reported for the Safety Population, which consisted of all subjects who received at least 1 application of study medication. There were 237 subjects in the SB206 QD group and 117 subjects in the Placebo group in the Safety Population.
Arm/Group | SB206 12% | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/237 | 0/117
Serious Adverse Events (participants affected / at risk) | 1/237 | 1/117
Other Adverse Events (participants affected / at risk) | 63/237 | 10/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB206 12% (N=237) | Placebo Comparator (N=117)
Cellulitis (Infections and infestations) | 1 (1) | 1 (3) — Moderate/unrelated/hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SB206 12% (N=237) | Placebo Comparator (N=117)
Application Site Pain (General disorders) | 37 | 0
Application site erythema (General disorders) | 26 | 0
Application site scar (General disorders) | 0 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must wait 18 months after the closeout of the trial at all Study sites or until the publication of the multi-site Sponsor results. The only restriction on PI publication after that time is that the sponsor can review results communications prior to public release and can request confidential or proprietary information be removed or can embargo communications regarding trial results for a period that is more than 90 days but less than 120 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT03927703/Prot_SAP_000.pdf